CLINICAL TRIAL: NCT00695747
Title: Intraocular Pressure Control Following One Site Versus Two Site Combined Phacoemulsification/IOL And Trabeculectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lahey Clinic (Other)
Responsible Party: Paul R. Cotran, M.D., Lahey Clinic, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 98-067
Record Dates: First submitted 2008-06-10; First posted 2008-06-12 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Glaucoma; Cataracts
Keywords: Glaucoma; Cataracts; Phacoemulsification(IOL); Trabeculectomy
MeSH Terms: conditions — Glaucoma; Cataract | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Standard 1 site Procedure using a fornix based incision, performed superiorly
- 2 (Experimental): 2 Site Combined Procedure
  Interventions: Procedure: 2 Site procedure- Phacoemulsification/IOL and Trabeculectomy

INTERVENTIONS:
Procedure: 2 Site procedure- Phacoemulsification/IOL and Trabeculectomy — 2 Site Combined Procedure: in which a temporal clear cornea approach would be used for the cataract/IOL part of the procedure, and immediately thereafter the superior limbus would be employed for a limbus-based trabeculectomy
  Other Names: Coexisting Cataract and glaucoma; Cateract; Glaucoma; Phacoemulsification/IOL; Trabeculectomy
  Arms: 2

SUMMARY:
The purpose of this study is to compare the safety & effectiveness of the two types of cataract and glaucoma surgeries. Results from this study may improve the surgical and post surgical management and long term management of patients with these conditions in the future

DETAILED DESCRIPTION:
The purpose of this study is to determine whether a Two-Site Technique for the Combined Procedure for subjects with coexisting visually significant glaucoma & cataracts will result in an improvement in IOP control in both the immediate and longer term postoperative period as compared with the currently Standard One Site surgical technique for both glaucoma and cataracts.

Research and data indicate that the success rate of the glaucoma part of this operation may be improved if the incision for the cataract part of the operation is separated from the drainage hole created for the glaucoma part, the constant drainage through this hole is what lowers the intraocular pressure after surgery. Using the Two-Site Combined procedure the glaucoma incision(drainage hole) will still be created superiorly, under the upper lid. The cataract incision will be moved to the temporal side of the eye ball, away from the drainage hole for the glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Meet the current criteria for combined procedure surgery:
* A visually significant cataract(ie: an opacification of the crystalline lens resulting in a reduction of visual performance affecting daily living
* Open angle or mixed mechanism glaucoma inadequately controlled on current therapy, or requiring two or more medications for control, or with advanced visual field and optic nerve damage.

Exclusion Criteria:

* Subjects with normal tension glaucoma(defined as those subjects in whom no IOPs greater than 21 mm Hg[preceding or during therapy]have been recorded)
* Subjects with uveitis
* Subjects with neovascular glaucoma
* Severe conjunctival inflammation or scarring
* Subjects who have had previous incisional ocular surgery in the same eye
* No subjects will have second eye operated on within 8 weeks of the first eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 1998-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Post-Op outcomes of IOP less than or equal to 16mm Hg without additional ocular hypotensive medications | Assessments made at 3 months post op, 3 month intervals for at least 2 years post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Paul R. Cotran, M.D., Principal Investigator — Lahey Clinic, Inc.
Locations (1):
- Lahey Clinic, Inc., Burlington, Massachusetts, United States

REFERENCES:
- [Background] Palmer SS. Mitomycin as adjunct chemotherapy with trabeculectomy. Ophthalmology. 1991 Mar;98(3):317-21. doi: 10.1016/s0161-6420(91)32293-0. PMID 2023752
- [Background] Shingleton BJ, Jacobson LM, Kuperwaser MC. Comparison of combined cataract and glaucoma surgery using planned extracapsular and phacoemulsification techniques. Ophthalmic Surg Lasers. 1995 Sep-Oct;26(5):414-9. PMID 8963855
- [Background] Gandolfi SA, Vecchi M. 5-fluorouracil in combined trabeculectomy and clear-cornea phacoemulsification with posterior chamber intraocular lens implantation. A one-year randomized, controlled clinical trial. Ophthalmology. 1997 Feb;104(2):181-6. doi: 10.1016/s0161-6420(97)30336-4. PMID 9052620
- [Background] Shin DH, Simone PA, Song MS, Reed SY, Juzych MS, Kim C, Hughes BA. Adjunctive subconjunctival mitomycin C in glaucoma triple procedure. Ophthalmology. 1995 Oct;102(10):1550-8. doi: 10.1016/s0161-6420(95)30832-9. PMID 9097805
- [Background] Joos KM, Bueche MJ, Palmberg PF, Feuer WJ, Grajewski AL. One-year follow-up results of combined mitomycin C trabeculectomy and extracapsular cataract extraction. Ophthalmology. 1995 Jan;102(1):76-83. doi: 10.1016/s0161-6420(95)31050-0. PMID 7831046
- [Background] Berestka JS, Brown SV. Limbus- versus fornix-based conjunctival flaps in combined phacoemulsification and mitomycin C trabeculectomy surgery. Ophthalmology. 1997 Feb;104(2):187-96. doi: 10.1016/s0161-6420(97)30335-2. PMID 9052621
- [Background] Scott IU, Greenfield DS, Schiffman J, Nicolela MT, Rueda JC, Tsai JC, Palmberg PF. Outcomes of primary trabeculectomy with the use of adjunctive mitomycin. Arch Ophthalmol. 1998 Mar;116(3):286-91. doi: 10.1001/archopht.116.3.286. PMID 9514480
- [Background] Parrish RK II, Folberg R. Wound healing in glaucoma surgery: In: Ritch R. Shields MB, Krupin T, eds. The Glaucomas 2nd ed. St. Louis: CV Mosby 1989, vol III, chap. 81